CLINICAL TRIAL: NCT00606411
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Determine the Efficacy and Safety of Topiramate in the Treatment of Sleep-Related Eating Disorder
Brief Title: Efficacy and Safety of Topiramate in the Treatment of Sleep-Related Eating Disorder
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, John Winkelman, MD, PhD, Associate Professor of Psychiatry, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MGH-2008P000662
Record Dates: First submitted 2008-01-22; First posted 2008-02-04 (Estimated); Results first posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Sleep-Related Eating Disorder
Keywords: Sleep-Related Eating Disorder; Topiramate; Parasomnia
MeSH Terms: conditions — Parasomnias | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topiramate (Active Comparator): Study medication arm, 25-300mg of Topiramate
  Interventions: Drug: Topiramate or Placebo
- Placebo (Placebo Comparator): Placebo arm of study, 25-300mg of sugar pill
  Interventions: Drug: Topiramate or Placebo

INTERVENTIONS:
Drug: Topiramate or Placebo — 25-300 mg tablets of topiramate and matching placebo, placed in blinded capsules
  Other Names: Brand Name: Topamax

SUMMARY:
The purpose of the study is to learn about the safety and effectiveness of oral (taken by mouth) topiramate in treating Sleep-Related Eating Disorder (SRED).

DETAILED DESCRIPTION:
This is a single center, 13-week, outpatient, randomized, double-blind, placebo-controlled, parallel group, pilot study of topiramate in subjects with Sleep-Related Eating Disorder (SRED). The primary objective of this study is to investigate the efficacy and safety of topiramate compared to placebo in the treatment of Sleep-Related Eating Disorder. SRED is a disorder that consists of out of control eating during the night with little or no awareness of the events. In this study we are comparing topiramate to placebo. A placebo is a pill that looks exactly like the study drug, but it does not have any active drug in it. Topamax (topiramate) is approved by the U.S. Food and Drug Administration (FDA) as a therapy for epilepsy, but topiramate has not been approved by the FDA for SRED.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65
* Diagnosis of SRED
* Must be able to swallow capsules and follow instructions

Exclusion Criteria:

* Women who are pregnant or lactating
* Other sleep disorders
* Kidney or Liver disease
* Night shift workers
* Previous history of Topiramate or Topamax use for any condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2018-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John W Winkelman, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Winkelman JW, Wipper B, Purks J, Mei L, Schoerning L. Topiramate reduces nocturnal eating in sleep-related eating disorder. Sleep. 2020 Sep 14;43(9):zsaa060. doi: 10.1093/sleep/zsaa060. PMID 32227216

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Topiramate | Placebo
Started | 16 | 18
Completed | 10 | 11
Not Completed | 6 | 7
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Adherence | 1 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 1 | 2
Not completed — Move out of state | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topiramate | Placebo | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (12) | 39.4 (12.1) | 39.5 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 3 | 6 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 14 | 15 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Number of nights eating per week [Mean (Standard Deviation); unit: percent of nights per week] | 74.7 (17.3) | 77 (17.2) | 75.2 (17.4)
Weight [Mean (Standard Deviation); unit: lbs] | 181.8 (38.5) | 188.2 (42.3) | 185.3 (40.1)
HbA1c [Mean (Standard Deviation); unit: percent glycohemoglobin/total hemoglobin] | 5.4 (0.2) | 5.3 (0.5) | 5.3 (0.4)
Average nightly total sleep time [Mean (Standard Deviation); unit: hours] | 7.0 (1.0) | 7.0 (1.1) | 7.0 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Frequency of Sleep-related Eating Episodes (Time Frame: Comparing Final Study Visit to Baseline)
Description: Frequency of sleep-related eating episodes was measured as the number of nights a participant had an episode within the previous two weeks. The change was measured by comparing the last study visit (by the participant) from to the baseline results.
Time Frame: every 2 weeks for 10 weeks
Population: One participant in the Topiramate group and one participant in the Placebo group were not analyzed due to being removed or withdrawing from the study prior to the collection of post-randomization data.
Measure: Mean (95% Confidence Interval); unit: change in % of nights eating per week
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 15 | 17
change in % of nights eating per week | -41.2 [-71.9 to -10.5] | -20.0 [-43.5 to 3.5]

2. Primary Outcome: The Clinician Global Impression (CGI) Scale
Description: The Clinician Global Impression (CGI) Scale is used by healthcare professionals to assess the overall severity of illness and change in a patient's condition over time. The scale ranges from 1 to 7, 1 being Very much improved and 7 being Very much worse. A participant with a score of 1 or 2 on the Clinician Global Impression scale was considered a "responder."
Time Frame: Day 1 (First Study Visit) to Day 63 (Final Study Visit) (assessed at last study visit)
Population: Two participants in the Topiramate group and three participants in the Placebo group were not analyzed due to being removed or withdrawing from the study prior to the end of treatment visit, where CGI is determined.
Measure: Number; unit: percentage responders
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 14 | 15
percentage responders | 71.4 | 26.7

3. Secondary Outcome: Body Weight
Description: The change in body weight in the study participants was calculated comparing the participant's last study visit to their baseline weight.
Time Frame: every other week for 10 weeks
Population: Two participants in the Topiramate group and four participants in the Placebo group were excluded from the analysis due to being removed or withdrawing from the study prior to the collection of this end-of-treatment datapoint.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 14 | 14
pounds | -8.5 (8.2) | 1.0 (5.3)

4. Secondary Outcome: HbA1c (%)
Description: Change in HbA1c levels from randomization to the end of follow-up.
Time Frame: Day 1 (First Study Visit) to Day 63 (Final Study Visit)
Population: Four participants in the Topiramate group and ten participants in the Placebo group were excluded from this analysis due to being removed or withdrawing from the study prior to the collection of this end of treatment data point.
Measure: Mean (95% Confidence Interval); unit: Change in percent HbA1c
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 12 | 8
Change in percent HbA1c | 0 [-0.1 to 0.1] | -0.2 [-0.4 to 0]

5. Secondary Outcome: Average Total Sleep Time (Hours)
Description: Average sleep time over the course of the previous two weeks, comparing end results to baseline.
Time Frame: Day 1 (First Study Visit) to Day 63 (Final Study Visit)
Population: Four participants in the Topiramate group and one participant in the Placebo group were excluded from the analysis due to being removed or withdrawing from the study prior to the collection of this end-of-treatment datapoint.
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 12 | 17
hours | 0.4 [-0.3 to 1.1] | 0.4 [-0.7 to 1.5]

6. Secondary Outcome: Sleep Quality (Visual Analogue Scale or VAS)
Description: Measured on visual analogue scale (VAS). VAS ranges were as follows: Sleep Quality; 0 = "Poorly" to 100 = "Great," Wakefulness; 0 = "Asleep/Not Awake" to 100 = "Fully Awake," Control; 0 = "No Control Over Eating" to 100 = "Full Control Over Eating," Memory; 0 = "No Memory of Eating" to 100 = "Fully Remember Eating". The change was calculated from baseline to the final study visit (day 63).
Time Frame: Day 1 (First Study Visit) to Day 63 (Final Study Visit)
Population: Two participants in the Topiramate group and two participants in the Placebo group were excluded from the analysis due to being removed or withdrawing from the study prior to the collection of this end-of-treatment datapoint.
Measure: Mean (Standard Deviation); unit: change in points on VAS (BL to day 63)
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 14 | 16
change in points on VAS (BL to day 63) | 3.0 (14.6) | -1.0 (17.0)

7. Secondary Outcome: The Patient Global Impression (PGI) Scale
Description: A participant with a score of 1 or 2 on the Patient Global Impression scale was considered a "responder."
Time Frame: Day 1 (First Study Visit) to Day 63 (Final Study Visit) (assessed at last study visit)
Population: Four participants in the Topiramate group and six participants in the Placebo group were excluded from the analysis due to being removed or withdrawing from the study prior to the collection of this end-of-treatment datapoint.
Measure: Number; unit: % Responders
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 12 | 12
% Responders | 75 | 16.7

ADVERSE EVENTS:
Time Frame: AE data collected over the course of 9-week titration period.
Arm/Group | Topiramate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/18
Other Adverse Events (participants affected / at risk) | 13/16 | 5/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Topiramate (N=16) | Placebo (N=18)
Paresthesia (Nervous system disorders) | 9 | 0
Dysgeusia (Nervous system disorders) | 5 | 0
Cognitive Dysfunction (General disorders) | 5 | 1
Daytime Tiredness (General disorders) | 5 | 3
Decreased Daytime Apetite (Metabolism and nutrition disorders) | 3 | 1
Dry Mouth (General disorders) | 3 | 0
Nausea (General disorders) | 1 | 0
Headache (General disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT00606411/Prot_SAP_000.pdf